CLINICAL TRIAL: NCT00728273
Title: Efficacy of Multiple Micronutrient Fortified Biscuits and Deworming on Reducing Anemia Prevalence, and Improving Micronutrient Status, Cognitive Function, and Growth in Vietnamese School Children
Brief Title: Efficacy of Multiple Micronutrient Fortified Biscuits and Deworming in Vietnamese School Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neys-van Hoogstraten Foundation, The Netherlands (Other)
Responsible Party: Principal Investigator: Dr. Pattanee Winichagoon, Ph.D., Associate Professor, Institute of Nutrition, Mahidol University, Nakhon Pathom, Thailand, 73170.
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Neys-code VT 188
Record Dates: First submitted 2008-07-30; First posted 2008-08-05 (Estimated); Last update posted 2008-12-04 (Estimated); Status verified 2008-11

CONDITIONS: Healthy
Keywords: Efficacy; Vietnam; school children; anemia; fortification; micronutrient
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- MMF (Experimental): multi-micronutrient-fortified biscuit plus placebo deworming-treatment
  Interventions: Dietary Supplement: worm treatment and multiple micronutrient fortified biscuits
- Alb (Experimental): placebo biscuit plus deworming treatment with Albendazole
  Interventions: Dietary Supplement: worm treatment and multiple micronutrient fortified biscuits
- MMF + Alb (Experimental): multiple micronutrient-fortified biscuits with deworming treatment with Albendazole
  Interventions: Dietary Supplement: worm treatment and multiple micronutrient fortified biscuits
- placebo (Placebo Comparator): placebo biscuit (non-fortified) and placebo deworming treatment
  Interventions: Dietary Supplement: worm treatment and multiple micronutrient fortified biscuits

INTERVENTIONS:
Dietary Supplement: worm treatment and multiple micronutrient fortified biscuits — A single dose of intestinal anthelminthic treatment as orange-flavored chewable tablets containing 400 mg Albendazole (Vidoca, Thephaco, Vietnam) was given. Deworming was repeated with Albendazole for all children at the end of the study (after 4 months).
  The composition and amount of nutrients in each serving of fortified biscuit were 6 mg iron, 5.6 mg zinc, 35µg iodine, 300 µg RAE vitamin A, 1.0 mg thiamin, 0.9 mg riboflavin, 1.1 mg vitamin B6, 10.5 mg NE niacin, 1.5 µg vitamin B12, 120 µg folic acid, 28 mg vitamin C, 150 mg calcium, 74 IU vitamin D, 40 mg magnesium, 6.8 µg selenium, 378 mg potassium, 70 mg phosphorus, 3.0 mg pantothenic acid, 2.8 µg vitamin E, 10 µg vitamin K and 18 µg biotin.
  Other Names: Vidoca (Thephaco, Vietnam)

SUMMARY:
The aim of this study is to identify the effect of a school-based food fortification intervention with multi-micronutrients with or without deworming to improve anemia, micronutrient status, cognitive function, health (morbidity and reinfestation rate) and growth (ponderal) in Vietnamese primary schoolchildren.

DETAILED DESCRIPTION:
Concurrent micronutrient deficiencies are prevalent in schoolchildren in Vietnam. These deficiencies not only lead to anemia, impair growth, increase susceptibility to infection, impair work capacity, but also impair cognitive development and impair learning ability. The risk of micronutrient deficiencies and anemia increases when individuals are exposed to intestinal helminth infections. Schoolchildren are a neglected group with regard to micronutrient interventions, and school programs afford an excellent opportunity to improve health of these groups. Food fortification with multi-micronutrients is a cost-effective and sustainable strategy, but is not yet implemented on a large scale in Vietnam. Furthermore, little is known about whether high prevalence of intestinal helminthic infection in schoolchildren limits the effect of fortification when this is not combined with regular de-worming.

ELIGIBILITY:
Inclusion Criteria:

* school children aged 6-8 years with written informed consent from parents/caregivers

Exclusion Criteria:

* hemoglobin concentrations < 80g/L
* chronic disease
* congenital abnormalities
* mental or severe physical handicap
* severe malnutrition
* obesity
* receiving deworming within the previous 6 mo

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 510 (Actual)
Dates: Start 2007-01; Primary Completion 2007-01 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of anemia, micronutrient status (iron, vitamin A, zinc, and iodine), and cognitive function (attention, IQ, concentration, and school achievement). | 4 months

SECONDARY OUTCOMES:
growth (especially weight), body composition (body fat) | 4 months
prevalence and incidence of infectious diseases such as diarrhea and respiratory infection over a 4-month period during the school feeding in | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Pattanee Winichagoon, PhD, Principal Investigator — Institute of Nutrition, Mahidol University, Nakhon Pathom, Thailand
Locations (1):
- Institute of Nutrition, Mahidol University, Nakhon Pathom, Thailand